CLINICAL TRIAL: NCT03274843
Title: Evaluation of the Improvement of Independence by the Resumption of a Significant Activity Such as a Cooking Workshop in Adult Patients With Stroke Benefiting From Traditional Rehabilitation
Acronym: EVIC-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC15_3021_EVIC-AVC
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with stroke (Experimental)
  Interventions: Other: Activity of everyday life

INTERVENTIONS:
Other: Activity of everyday life — Kitchen workshop

SUMMARY:
A non-randomized, monocentric, pilot study comparing the level of independence for each individual with significant resumption of activity in adult patients with stroke

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Primary stroke or recurrence on stroke having no previous sequelae
* Stroke older than 3 weeks
* Ability to understand treatment and sufficient motivation
* Problem Activity Indicated in CMOP (Canadian Measure of Occupational Performance)
* Barthel Index > 60
* Patient who received oral and written information about the protocol and who did not show opposition to participate in the study

Exclusion Criteria:

* Dermatological pathology with wounds on the unhealed upper limbs
* Patient in contact and droplet isolation
* A psychiatric history requiring hospitalization in specialized settings for more than 2 months
* Any condition that may limit participation or interfere with analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of independence in a population of adult patients with stroke having participated in cooking workshop at week 3 | Day 0, Week 3
  Evaluation of independence by Functional Independence Measure score

SECONDARY OUTCOMES:
Evaluation of the patient's quality of life | Day 0, Week 3
  Evaluation of the patient's quality of life by the Medical Outcome Study (MOS)Short Form (SF-36 ) questionnaire
Evaluation of the patient's self-esteem | Day 0, Week 3
  Evaluation of the patient's self-esteem by Rosenberg Self Estimate Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No